CLINICAL TRIAL: NCT00799045
Title: Clopidogrel On Top of Aspirin For the Prevention of New Onset Migraine Headache Occurrence Following Transcatheter Closure of Atrial Septal Defects: A Prospective Randomized Trial (the CANOA Study)
Brief Title: Clopidogrel For the Prevention of New Onset Migraine Headache Following Transcatheter Closure of Atrial Septal Defects
Acronym: CANOA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Sanofi (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLOPI_L_03563
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Migraine
Keywords: Migraine; atrial septal defects; transcatheter; clopidogrel
MeSH Terms: conditions — Migraine Disorders; Heart Septal Defects, Atrial | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin + clopidogrel (Experimental): Aspirin (80 mg/day) + clopidogrel (75 mg/day) for 3 months following ASD closure.
  Interventions: Drug: Clopidogrel
- Aspirin (Active Comparator): Aspirin (80 mg/day) for 3 months following ASD closure.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Patients will be randomized either to aspirin (80 mg/day) or aspirin (80 mg/day) + clopidogrel (75 mg/day) for 3 months following ASD closure.
  Other Names: Clopidogrel (Plavix)

SUMMARY:
The addition of clopidogrel on top of aspirin may reduce the occurrence of new-onset migraine headache episodes following transcatheter ASD closure.

DETAILED DESCRIPTION:
The objective is to evaluate the incidence and severity of new-onset migraine headache episodes following transcatheter ASD closure in patients treated with aspirin alone compared to those on aspirin + clopidogrel therapy as antithrombotic treatment after the procedure.

This is a prospective, randomized, double blind, multicenter study, including patients with no previous history of migraine attacks who have been diagnosed with an ASD and for whom transcatheter ASD closure has been clinically indicated. Patients will be randomized either to aspirin (80 mg/day) or aspirin (80 mg/day) + clopidogrel (75 mg/day) for 3 months following ASD closure. The occurrence and severity of migraine headaches will be evaluated by a neurologist using a structured headache questionnaire at 1 month and 3 months following ASD closure. An additional 6 month and 1 year follow-up evaluation will be exploratory according to local feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year old undergoing transcatheter ASD closure with the Amplatzer Septal Occluder device (AGA medical Corp., MN, USA).
* Female subjects must be post-menopausal, surgically sterile, or using an effective method of birth control.
* Signed an informed consent document.

Exclusion Criteria:

* Allergy or intolerance to any of the antithrombotic drugs (aspirin, clopidogrel) used in the study.
* Need for anticoagulation therapy.
* Use of ASD closure devices other than the Amplatzer Septal Occluder device.
* History of migraine headaches (based on migraine headache questionnaire).
* Refusal to sign the informed consent.
* Pregnancy or breast-feeding or planning to become pregnant during the study.
* Previous stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-10; Primary Completion 2015-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean number of monthly migraine days per patient within the 3 months following transcatheter ASD closure. | 3 months

SECONDARY OUTCOMES:
Severity of migraine attacks following ASD closure as evaluated by the intensity of migraine episodes and the Migraine Disability Assessment (MIDAS) questionnaire at 3-month follow-up after ASD closure. | 3 months
Incidence of bleeding complications at 3-month follow-up. | 3 months
Percentage of patients with new-onset migraine attacks. | 3 months
Time to first migraine episode. | 3 months
Percentage of patients with migraine headaches at 6-month and 1-year follow-up (exploratory only according to local feasibility). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodes-Cabau, MD, Principal Investigator — Hopital Laval
Locations (1):
- Hopital Laval, Québec, Canada

REFERENCES:
- [Derived] Wintzer-Wehekind J, Horlick E, Ibrahim R, Cheema AN, Labinaz M, Nadeem N, Osten M, Cote M, Marsal JR, Rivest D, Marrero A, Houde C, Rodes-Cabau J. Effect of Clopidogrel and Aspirin vs Aspirin Alone on Migraine Headaches After Transcatheter Atrial Septal Defect Closure: One-Year Results of the CANOA Randomized Clinical Trial. JAMA Cardiol. 2021 Feb 1;6(2):209-213. doi: 10.1001/jamacardio.2020.4297. PMID 32965476
- [Derived] Rodes-Cabau J, Horlick E, Ibrahim R, Cheema AN, Labinaz M, Nadeem N, Osten M, Cote M, Marsal JR, Rivest D, Marrero A, Houde C. Effect of Clopidogrel and Aspirin vs Aspirin Alone on Migraine Headaches After Transcatheter Atrial Septal Defect Closure: The CANOA Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2147-54. doi: 10.1001/jama.2015.13919. PMID 26551304